CLINICAL TRIAL: NCT07217990
Title: Neoadjuvant Complete Response Customized Treatment Approach for Definitive Management of Breast Cancer
Acronym: NoCUT-BC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Principal Investigator, Sachin Jhawar, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-25103; NCI-2025-07434 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Neoadjuvant Therapy; Radiotherapy; Magnetic Resonance Spectroscopy; Mastectomy, Segmental; Mastectomy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (eeCR, non-surgical) (Experimental): Patients will receive standard of care (SOC) neoadjuvant chemotherapy and will be evaluated for enhanced clinical complete response (ecCR) after treatment. Participants who achieve an ecCR will be placed in the non-surgical arm. Participants will receive radiation therapy and routine and additional screening MRIs during follow up.
  Interventions: Drug: Neoadjuvant Chemotherapy; Radiation: Radiation Therapy; Procedure: MRI; Procedure: Biopsy; Procedure: Biospecimen collection
- Arm B (non-eeCR, surgical) (Experimental): Patients will receive standard of care (SOC) neoadjuvant chemotherapy and will be evaluated for enhanced clinical complete response (ecCR) after treatment. Participants who do not achieve an ecCR will be placed in the surgical arm. Participants will undergo a lumpectomy or mastectomy, receive radiation therapy, and routine follow-up.
  Interventions: Drug: Neoadjuvant Chemotherapy; Radiation: Radiation Therapy; Procedure: MRI; Procedure: Breast Cancer Surgery; Procedure: Biopsy; Procedure: Biospecimen collection

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Participants will receive standard of care neoadjuvant chemotherapy
Radiation: Radiation Therapy — Radiotherapy simulation parameters will be at the discretion of the treating physician to account for the patient's body habitus, tumor bed location, and tolerability of the prone or supine positions, however, the recommended approach will be whole-breast RT (WBRT) in the prone position, for cT1-3 N0 patients who achieve ecCR. For cT1-2 N1 patients who achieve ecCR WBRT with nodal inclusion and lymph node boost will be performed in the supine position.
  Other Names: Radiotherapy
Procedure: MRI — Participants will undergo MRI
  Other Names: Magnetic Resonance Imaging
Procedure: Breast Cancer Surgery — Participants will undergo surgery to treat their breast cancer. Either a lumpectomy or a mastectomy will be performed.
  Other Names: Lumpectomy; Mastectomy
  Arms: Arm B (non-eeCR, surgical)
Procedure: Biopsy — Participants undergo biopsy
Procedure: Biospecimen collection — Participants undergo blood and plasma collection

SUMMARY:
This study will evaluate the efficacy and non-inferiority of a non-surgical approach for the treatment of patients with locally advanced breast cancer.

DETAILED DESCRIPTION:
Primary Objective: To determine if a non-surgical approach to breast cancer patients with an exceptional response to NAC leads to similar recurrence rates compared to standard of care (SOC).

Exploratory Objectives

1. To study personalized predictive biomarkers of response to chemotherapy and predictors of residual disease from tumor samples and circulating biomarkers.
2. To validate our internally developed deep learning model to predict pathological complete response (pCR) postNAC in breast cancer patients.

Outline: This is a phase II trial that will accrue up to 84 participants. Patients will receive standard of care (SOC) neoadjuvant chemotherapy and will be evaluated for enhanced clinical complete response (ecCR) after treatment. The ecCR will be evaluated using a trimodal approach, which includes the use to Magnetic Resonance Imaging (MRI), image-guided biopsy, and circulating tumor DNA (ctDNA) analysis. Participants who achieve an ecCR will be placed in the non-surgical arm (Arm A), while those who do not achieve an ecCR will be placed in the surgical arm (Arm B).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older
4. Early-stage breast cancer diagnosis (cT1-3 N0 or cT1-2 N1) and a Human Epidermal Receptor 2 (HER2)-positive or triple negative breast cancer (TNBC) tumor molecular subtype
5. Planning to receive neoadjuvant chemotherapy (NAC) and radiation therapy (RT)

Exclusion Criteria:

1. Pregnancy or lactation
2. Inmate or prisoner
3. Treatment with an investigational drug or other intervention throughout their breast cancer treatment
4. Patients with skin involvement and/or distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Rate | At 12 months
  The study endpoints of disease-free rate and locoregional control will be determined in patient follow up by utilizing MRIs, annual mammograms and clinical assessments in conjunction with ctDNA status.

SECONDARY OUTCOMES:
Locoregional control | At 2, 3 and 5 years
  The study endpoints of disease-free rate and locoregional control will be determined in patient follow up by utilizing MRIs, annual mammograms and clinical assessments in conjunction with ctDNA status.
Disease-free survival | Up to 5 years
  Survival analysis will be conducted for time to event data, and the disease control or survival rate at specific times will be estimated based on the survival analysis along with the 95% CI.
Treatment related adverse events | Up to 5 years
  Toxicities will be recorded using CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Jhawar, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu